CLINICAL TRIAL: NCT05896553
Title: Effects of Oxytocin on the Functional Architecture of the Brain Before and After Prolonged Naturalistic Fear Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-BAM-08
Record Dates: First submitted 2023-05-29; First posted 2023-06-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy
Keywords: Oxytoxin; Fear; fMRI; Functional Connectivity

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled double-blind between-subject design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytoxin group (Experimental): Drug: intranasal Oxytocin(24IU)
  Interventions: Drug: intranasal Oxytocin(24IU)
- Placebo group (Placebo Comparator): Drug: intranasal Placebo
  Interventions: Drug: intranasal Placebo

INTERVENTIONS:
Drug: intranasal Oxytocin(24IU) — Administration of intranasal Oxytocin(24IU)
  Arms: Oxytoxin group
Drug: intranasal Placebo — Administration of intranasal Placebo
  Arms: Placebo group

SUMMARY:
The main aim of the pharmacological resting-state fMRI study is to investigate the modulatory effects of intranasal Oxytocin (24IU) on task and intrinsic functional connectivity before and after prolonged exposure to naturalistic fear induction via a movie.

DETAILED DESCRIPTION:
In a double-blind placebo-controlled between-subject experimental design, 60 adult male subjects will be randomly allocated to either receive intranasal Oxytocin (24IU, n= 30) or intranasal placebo (nasal spray administration without oxytocin, n = 30). Following treatment administration subjects will undergo a resting state functional magnetic resonance imaging (fMRI) assessment (8min) and next watch a long fear-inducing (horror) movie (10min) followed by a resting state fMRI assessment (8min). Effects of treatment on subjective experience will be assessed using 1-9 Likert scales assessing subjective fear, emotional arousal and escape. Ratings will be acquired before the start of the experiment, after the movie and at the end of the experiment. Participants will undergo screening for psychopathological and emotional states before treatment. Together with a randomized assignment to the treatment groups, this will allow controlling for confounding between-group differences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without past or current psychiatric or neurological disorders
* Right-handedness
* Normal or corrected-normal version

Exclusion Criteria:

* History of head injury
* Medical or psychiatric illness
* Hypertension
* General cardio-vascular alteration or diseases
* Allergy against medications
* Visual or motor impairments
* Claustrophobia
* Drug addiction
* Nicotine dependence
* FMRI contradictions

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Functional connectivity during the resting state between brain systems involved in emotional processing. | Change between the time windows 72-80 minutes (before emotion induction) and 90-98 minutes (after emotion induction) following treatment
  1.During the 8min resting state before and after the movie clips the intrinsic connectivity of the brain will be assessed. The intrinsic connectivity will be computed as temporal correlation between spatially remote neurophysiological events, expressed as deviation from statistical independence across these events in distributed neuronal groups and areas. Effects of Oxytocin on the intrinsic architecture of the brain will be examined by comparing the Oxytocin- and Placebo- treated groups.

SECONDARY OUTCOMES:
Functional and dynamic connectivity during the movie clip will be examined during the fear-induction period (10min movie clip). | 80 minutes to 90 minutes after treatment
  Effects of treatment on dynamic functional connectivity during the fear clip watching phase will be examined by comparing dynamic functional connectivity indices between the Oxytoxin- and Placebo-treated group.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Dr., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No